CLINICAL TRIAL: NCT01690377
Title: Plasmacytoid Dendritic Cells in Vaccination of Stage IV Melanoma Patients: a Phase I Study
Brief Title: Natural Dendritic Cell Vaccines in Metastatic Melanoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-093; KWF 2004-3127
Record Dates: First submitted 2008-02-05; First posted 2012-09-21 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Melanoma
Keywords: Dendritic Cells
MeSH Terms: conditions — Melanoma | interventions — phosducin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PDC or myDC
  Interventions: Biological: PDC or myDC

INTERVENTIONS:
Biological: PDC or myDC — PDC or myDC; first patient 0.3 * 10E6 PDC; second and third 1 * 10E6 PDC; fourth and fifth 3 * 10E6 PDC.

SUMMARY:
Dendritic cells (DCs) are the professional antigen-presenting cells of the immune system. As such they are currently used in clinical vaccination protocols in cancer patients, and both immunological and clinical responses have been observed. Several subsets of dendritic cells have been characterized in the peripheral blood. One such subset is referred to as plasmacytoid dendritic cells (PDC), another as myeloid dendritic cells (myDC). To date PDC and myDC have not been evaluated for their capability to induce anti-tumor immune responses in patients. For this reason the investigators will perform a safety and efficacy study with PDC and myDC in stage IV melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV melanoma according to the 2001 AJCC criteria. Limited tumor burden; LDH < 2x upper limit of normal
* Histological proof of cutaneous melanoma
* Melanoma expressing tyrosinase and/or gp100 (approximately 20% of cells or more determined by immunohistochemistry staining)
* HLA Type A2
* WBC > 3.0 * 10E9/l, lymphocytes > 0.8 * 10E9/l, platelets > 100 * 10E9/l, serum creatinine < 150 umol/l, serum bilirubin < 25 umol/l, normal liver function
* Expected adequacy of follow up
* Written informed consent

Exclusion Criteria:

* autoimmune disorders, concomitant use of immunosuppressive drugs
* serious concomitant disease, serious active infections, other malignancy in the past 5 years with the exception of curatively treated carcinoma in-situ of the cervix/squamous cell carcinoma of the skin
* known allergy to shell fish (vaccine contains KLH)
* pregnancy or lactation
* clinical signs of CNS metastases, in patients with a clinical suspicion of CNS metastases, a CT scan of the brain should be performed to exclude this
* prior chemotherapy, immunotherapy, or radiotherapy within three months before planned vaccination is allowed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
intervention-related toxicity | Within the first 6 months
  all adverse events within a time frame of 3 weeks after the last vaccination will be scored according to Common Terminology Criteria for Adverse Events (CTCAE)Version 4.0

SECONDARY OUTCOMES:
Immunological response | Within the first year
  The immunological response will be determined by tetramer sampling of skin-test derived lymphocyte cultures and peripheral blood after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: C J A Punt, MD, PhD, Principal Investigator — Radboud University Medical Center; C G Figdor, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre / Nijmegen Centre for Molecular Life Sciences
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands